CLINICAL TRIAL: NCT03277846
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Safety and Efficacy of Nexalin Electrical Brain Stimulation for the Treatment of Depression in Patients Referred to Electro-Convulsive Therapy
Brief Title: The Safety and Efficacy of Nexalin Trans-cranial Electrical Stimulation Stimulation for the Treatment of Depression
Acronym: TES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Carrier Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 824349
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Results first posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: A 2x2 factor Randomized Controlled Trial with block randomization
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants and investigators are blind to condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (4):
- Accept ECT - TES (Experimental): Accept ECT where subject is randomized to TES
  Interventions: Device: Nexalin Based Trans-Cranial Electrical Stimulation
- Accept ECT - SHAM (Placebo Comparator): Accept ECT where subject is randomized to a SHAM condition
  Interventions: Device: Nexalin Based Trans-Cranial Electrical Stimulation
- Reject ECT - TES (Experimental): Reject ECT where subject is randomized to TES
  Interventions: Device: Nexalin Based Trans-Cranial Electrical Stimulation
- Reject ECT - SHAM (Placebo Comparator): Reject ECT where subject is randomized to SHAM
  Interventions: Device: Nexalin Based Trans-Cranial Electrical Stimulation

INTERVENTIONS:
Device: Nexalin Based Trans-Cranial Electrical Stimulation — The Nexalin device, FDA clearance (501K=K024377, Classification: Stimulator, Cranial Electrotherapy: CFR 882. 5800: U.S. Patent #6904322B2), produces a square waveform that provides trans-cranial electrical stimulation to the brain delivered at a frequency of 77.5 Hz at 0 to 4 mA peak current.
  Other Names: TES

SUMMARY:
The purpose of this research study is to determine whether Nexalin Trans-Cranial Electrical Stimulation (TES) is an effective treatment for depression among patients who are candidates for ECT. A secondary aim to assess whether Nexalin can be used as an alternative to ECT. Although Nexalin has been approved for use in the US, using Nexalin to treat depression in this way is investigational and experimental. If Nexalin is found to be an alternative to ECT, it could offer a safer treatment for depression with less side-effects and a lower cost.

!!! NOTE !!! Post Script / Post Study. The ECT arm (profiling subjects as ECT accepters vs. rejecters) was dropped owing to site objections by referring clinicians. Accordingly, the study was framed as a simple comparison between TES and SHAM TES.

DETAILED DESCRIPTION:
A 2x2 factor Randomized Controlled Trial with block randomization. Inpatient subjects at the Carrier Clinic who are referred for ECT will be recruited, typed regarding their acceptance of ECT, and randomized to either treatment with TES or to a Sham condition. Treatment non-responders in either condition will continue as in patients at the Carrier Clinic until they reach acceptable levels of functioning to be discharged.

ELIGIBILITY:
Inclusion Criteria:

1. In-patients at the Carrier Clinic
2. Adults over age 18 and under age 65
3. Able to speak, read and write fluently in English, assessed by the study coordinator at Carrier Clinic
4. Screened Negative for alcohol abuse and/or dependence
5. Able to provide informed consent, assessed by the study coordinator at Carrier Clinic
6. Referred for ECT
7. Not currently taking hypnotics or be prescribed hypnotics during the Nexalin trial
8. Not pregnant or intending to become pregnant during the study
9. Committed to completion of the study

Exclusion Criteria: Medically or psychiatrically unstable, where the severity of the illness prohibits the subject from engaging in study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-05-17 (Actual); Study Completion 2018-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L Perlis, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Carrier Clinic, Belle Mead, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data will be shared with our collaborators at Nexalin and Carrier Clinic.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: with 6-18 months
Access Criteria: Only our direct collaborators.

REFERENCES:
- [Background] Bestmann S, Walsh V. Transcranial electrical stimulation. Curr Biol. 2017 Dec 4;27(23):R1258-R1262. doi: 10.1016/j.cub.2017.11.001. PMID 29207262
- [Background] Antal A, Alekseichuk I, Bikson M, Brockmoller J, Brunoni AR, Chen R, Cohen LG, Dowthwaite G, Ellrich J, Floel A, Fregni F, George MS, Hamilton R, Haueisen J, Herrmann CS, Hummel FC, Lefaucheur JP, Liebetanz D, Loo CK, McCaig CD, Miniussi C, Miranda PC, Moliadze V, Nitsche MA, Nowak R, Padberg F, Pascual-Leone A, Poppendieck W, Priori A, Rossi S, Rossini PM, Rothwell J, Rueger MA, Ruffini G, Schellhorn K, Siebner HR, Ugawa Y, Wexler A, Ziemann U, Hallett M, Paulus W. Low intensity transcranial electric stimulation: Safety, ethical, legal regulatory and application guidelines. Clin Neurophysiol. 2017 Sep;128(9):1774-1809. doi: 10.1016/j.clinph.2017.06.001. Epub 2017 Jun 19. PMID 28709880
- [Background] Yavari F, Jamil A, Mosayebi Samani M, Vidor LP, Nitsche MA. Basic and functional effects of transcranial Electrical Stimulation (tES)-An introduction. Neurosci Biobehav Rev. 2018 Feb;85:81-92. doi: 10.1016/j.neubiorev.2017.06.015. Epub 2017 Jul 6. PMID 28688701

RESULTS

PARTICIPANT FLOW:
Groups:
- Transcranial Electrical Stimulation (Active): All subjects get active treatment with Transcranial Electrical Stimulation
- TES SHAM: All subjects get SHAM treatment with TES
Period: Overall Study
Arm/Group | Transcranial Electrical Stimulation (Active) | TES SHAM
Started | 50 | 51
Completed | 38 | 40
Not Completed | 12 | 11
Not completed — Inpatient stay too brief | 12 | 11

BASELINE CHARACTERISTICS:
Groups:
- Transcranial Electrical Stimulation: Transcranial Electrical Stimulation (TES). Active Treatment.
- SHAM -TES: Sham/placebo condition
- Total: Total of all reporting groups
Arm/Group | Transcranial Electrical Stimulation | SHAM -TES | Total
Number analyzed (Participants) | 50 | 51 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 51 | 101
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (2.4) | 35.9 (2.3) | 34.2 (2.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 30 | 31 | 61
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 35 | 32 | 67
  African American | 3 | 0 | 3
  Asian | 0 | 1 | 1
  Native American | 0 | 1 | 1
  Multi-Racial | 0 | 2 | 2
  Hispanic | 4 | 5 | 9
  Unknown | 8 | 10 | 18
Region of Enrollment [Number; unit: participants]
  United States | 50 | 51 | 101

OUTCOME MEASURES:

1. Primary Outcome: Treatment Response
Description: Percent responders to TES treatment and Sham TES (50% reduction or a score below 10 on the PHQ-9). The PHQ-9 is a 9 item scale, where each item ranges from 0 to 3. Zero represents "not at all" and 3 represents "nearly every day". The scale ranges from 0-27. We used percent change (from admission to "ex-take") as a our metric.
Time Frame: 1-2 weeks
Population: 101 were enrolled. 78 subjects were in study for the minimum time / minimum number of treatments and provided the full compliment of data.
Measure: Count of Participants; unit: Participants
Groups:
- Transcranial Electrical Stimulation: Transcranial Electrical Stimulation (Active Tx)
- TES-SHAM: SHAM treatment (no current). Otherwise procedures identical.
Arm/Group | Transcranial Electrical Stimulation | TES-SHAM
Number analyzed (Participants) | 38 | 40
Participants | 28 | 29

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Transcranial Electrical Stimulation: TES = Transcranial Electrical Stimulation (active treatment)
- SHAM-TES: TES. No current. Procedures were otherwise identical between conditions
Arm/Group | Transcranial Electrical Stimulation | SHAM-TES
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/51
Other Adverse Events (participants affected / at risk) | 0/50 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/46/NCT03277846/Prot_SAP_000.pdf